CLINICAL TRIAL: NCT06807528
Title: Intermittent Fasting as an Anti-inflammatory Strategy for the Treatment of Depression in Spinal Cord Injury
Brief Title: Intermittent Fasting for Inflammation and Depression in Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15564
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injury; Depression - Major Depressive Disorder
Keywords: spinal cord injury; inflammation; depression; intermittent fasting
MeSH Terms: conditions — Spinal Cord Injuries; Inflammation; Depression; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Eligible participants who consent to study participation will be randomized to one of two groups: intermittent fasting + behavioral support techniques or intermittent fasting only. Each group will undergo 8-weeks of the respective treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting + Behavioral Support Strategies (Experimental): The intermittent fasting + behavioral strategies arm will follow a 16:8 protocol whereby they will be asked to fast for 16 hours per day and allowed to eat ad-libitum for the remaining 8 hours. This arm will also receive behavioral strategies including education, ongoing tailored feedback and encouragement, self monitoring tools, and goal setting will be used to help participants adhere to the fasting protocol. These techniques will be implemented via weekly phone calls to allow for coaching (e.g. barrier identification, strategies/action planning to overcome barriers, goal setting) as well as a smartphone app
  Interventions: Behavioral: Intermittent fasting; Behavioral: Behavioral Support Strategies
- Intermittent Fasting Only (Active Comparator): Participants allocated to the intermittent fasting only group will undergo the same 16:8 intermittent fasting protocol, however, they will not be provided with behavioral strategies via phone calls or the smart phone application. Weekly phone calls will be performed only for the purposes of assessing adherence, tracking adverse events, and ensuring participant safety.
  Interventions: Behavioral: Intermittent fasting

INTERVENTIONS:
Behavioral: Intermittent fasting — Participants will follow a 16:8 protocol whereby they will be asked to fast for 16 hours per day and allowed to eat ad-libitum for the remaining 8 hours. While (for feasibility purposes) it will be a requirement that the fasting period include time spent asleep, participants will be allowed some degree of flexibility in the start and end time of their fasting period. This will be performed in order to accommodate participant preferences (sleeping/eating/medication schedules) as best as possible and provide a sense of autonomy. During the non-fasting hours, participants will be permitted to eat ad libitum.
Behavioral: Behavioral Support Strategies — Evidence-based self regulatory health behaviour support techniques including education, ongoing tailored feedback and encouragement, self monitoring tools, and goal setting will be used to help participants adhere to the fasting protocol. These techniques will be implemented via weekly phone calls to allow for coaching (e.g. barrier identification, strategies/action planning to overcome barriers, goal setting) as well as a smartphone app. The smartphone application will provide information pertaining to intermittent fasting including lay summaries of clinical trials as well as infographics related to healthy eating for the ad-libitum eating periods. Tips for healthy eating on a budget and adhering to an intermittent fasting protocol will also be provided. The smartphone app will also feature intermittent fasting start and stop time reminders, hydration reminders, and the ability to set one's individualized fasting schedule and record actual daily fasting windows.
  Arms: Intermittent Fasting + Behavioral Support Strategies

SUMMARY:
Depression and chronic inflammation are common problems for people with spinal cord injury (SCI). Inflammation has been shown to influence depression which may make it an important treatment target. Previous studies have shown that changes in diet and exercise can affect this pathway and improve symptoms of depression in SCI patients. However, following these interventions long-term can be difficult.

Intermittent fasting is a way of eating that involves fasting for a certain period of time and then eating normally. It has been shown to reduce inflammation and improve mood in able-bodied people, but its unknown if it can help people with depression and chronic inflammation, such as those with SCI. As intermittent fasting is a simple, easier to follow strategy than a diet it may be a more feasible long-term strategy. In addition, certain behavioural techniques such education, encouragement, and self monitoring may further help. This study aims to find out if intermittent fasting + support can be a helpful and simpler treatment for depression in SCI patients.

In this study, 32 individuals with SCI who have depression will be invited to be randomly assigned to either try intermittent fasting + support or intermittent fasting alone. Both groups will fast for 16 hours per day for 8-weeks but only the supported group will receive behaviour techniques. Measurements will be taken prior to starting the interventions and after completing the interventions to assess for any changes in depression. Adherence, safety and inflammation will also be assessed.

By the end of the study, the investigators hope that intermittent fasting can help safely reduce symptoms of depression and inflammation in people with SCI. The investigators also hope to find that additional behavior support further helps people adhere. This may provide a simple, easy to follow, and cost-free treatment for depression and inflammation in people with SCI.

DETAILED DESCRIPTION:
Background: Depression and chronic inflammation are highly prevalent among individuals with spinal cord injury (SCI). Selective serotonin reuptake inhibitors (SSRIs) are the most prominently prescribed treatment strategy. While SSRIs can provide alleviation of symptoms for some patients, they are also associated with side-effects, and high rates of ineffectiveness/relapse. Due to the shortcomings of current treatments, it is critical to better understand factors which contribute to depressive symptoms and explore novel treatment modalities to improve outcomes for individuals with SCI and depression. Growing evidence suggests chronic inflammation plays a substantial role in the development of depression. Prior research from our lab has demonstrated this in SCI, as well as the efficacy of anti-inflammatory diets and exercise as treatments. However, adherence to these interventions over the long-term is challenging. Intermittent fasting (IF) has been shown to induce anti-inflammatory and anti-depressant effects in able-bodied individuals, and may be less burdensome, but its impact has not been evaluated in SCI. Further, behavioural support techniques such as education, ongoing tailored feedback and encouragement, self monitoring tools, and goal setting may help to further facilitate adherence to this less burdensome intervention strategy making it a more viable treatment long-term treatment option.

Objective/Hypothesis: The overall objective of this pilot study is to assess whether intermittent fasting combined with behavioral support techniques can provide a safe and feasible means of improving symptoms of depression in individuals with spinal cord injury (SCI) in comparison to an intermittent fasting only condition and explore the underlying mechanisms of action. This pilot will provide effect sizes to allow for a sample size calculation, and will assess the utility of implementing behavioral support techniques for a future larger scale RCT.

Methods: An RCT will be conducted involving 32 participants with mild to moderate depression recruited from the SCI outpatient program at Parkwood Institute. Participants will be randomly assigned to either the IF + support group or IF only group. The IF intervention will be performed by both groups over a period of 8-weeks whereby participants will fast daily (16-hour fast / 8-hour ad-libitum). The IF + support group will be provided with a smartphone app to provide behavioural support techniques, while the IF only group will not receive additional support. Outcome measures will be assessed at baseline and post intervention. The primary outcome measures will be changes in symptoms of depression and adherence to the intervention. Secondary outcomes will include safety, and change in inflammation and related pathways.

Significance: IF may provide a safe and feasible intervention to improve symptoms of depression following SCI. The addition of simple behavioral support techniques may enhance adherence further. The low burden and cost-free nature of this intervention may make it a more suitable long-term ant-inflammatory treatment strategy for depression for individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic (≥1 year post) SCI of any level or severity
2. 18 years of age or older
3. mild to moderate scores of depression based on the Structured Clinical Interview for DSM-5 (SCID) by clinical psychologist
4. stable dose of depression medications

Exclusion Criteria:

1. currently using anti-inflammatory medications
2. variable dosages of depression / anxiety medications
3. currently using anticoagulant medications
4. people with diabetes
5. women who are pregnant or attempting to become pregnant
6. current wound/infection
7. people with suicidal ideation
8. history of eating disorder
9. prior diagnosis of cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Symptoms of Depression | 8 weeks
  This study will assess changes in symptoms of depression (over 8-weeks) in response to the intermittent fasting + behavioral support techniques condition compared to an intermittent fasting only condition as measured by the patient health questionnaire-9 (PHQ-9).
  The PHQ-9 has been shown to be a valid assessment for major depressive disorder in individuals with SCI. The PHQ-9 is a 9-item questionnaire with items pertaining to feelings over the previous 2-weeks. Each item is scored on a scale from 0 ("not at all") to 3 ("nearly every day") with total scores allowing for assessment of depression severity. A score ranging from 0-4 suggests "none-minimal" depression severity, 5-9 suggests mild depression severity, 10-14 suggests moderate depression severity, 15-19 suggests moderately severe depression severity, and 20-27 suggests severe depression severity. A PHQ-9 score ≥ 10 has a sensitivity of 88% and a specificity of 88% for major depression.
Program Adherence Rates | 8 weeks
  Adherence will be assessed to examine how well participants in the intermittent fasting + behavioral support techniques condition adheres to the protocol compared to the intermittent fasting only condition. Adherence will be assessed based on self-reported eating times to determine the number of days participants in each group successfully adhered to the fasting condition. Specifically, days where participants performed the full 16 hour fasting window will be considered 'Adherent'. Days where participants do not perform the full 16 hour fasting window will be considered "Non-adherent'. Daily adherence percentage will be calculated based on the number of days participants were adherent divided by the total number of days of the intervention multiplied by 100.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events During Intervention | 8 weeks
  Safety of the intermittent fasting intervention will be assessed by evaluating the presence of any adverse events across all participants. Data pertaining to safety will be collected by the study team on a weekly basis during the weekly follow-up calls. Any incidence of treatment-emergent adverse events during the intervention will be recorded during these phone calls as well as at the final in-person visit. A description of the adverse event, severity of the adverse event, number of events, and total number of participants affected by each type of event will be recorded.
Anxiety | 8 weeks
  This study will assess changes in symptoms of anxiety (over 8-weeks) in response to the intermittent fasting + behavioral support techniques condition compared to the intermittent fasting only condition as measured by clinical assessment using the Generalized Anxiety Disorder-7 (GAD-7).
  The GAD-7 reflects symptoms of anxiety and respondents are asked to rate how often they have been "bothered" by these symptoms in the last two weeks on a scale from 0 (never) up to 3 (nearly every day). The items also provide a severity score from 0 - 21. Scores can be grouped as follows: ≤5 = no anxiety; 6-9 = mild anxiety; 10-14 = moderate anxiety, and ≥15 = severe anxiety.
Change in Plasma Cytokines | 8 weeks
  Blood samples (10ml) will be collected by a certified nurse/phlebotomist for the quantification of plasma cytokines (pg/ml) at baseline and 8-weeks (post intervention). Plasma concentrations of the pro-inflammatory cytokines tumour necrosis factor-alpha (TNF-α), C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-1 beta (IL-1β), and interferon-gamma (IFN-y) will be quantified using 32x4 simple plex multianalyte cartridge for the Ella automated immunoassay system (ProteinSimple, San Jose, California). Each of the cytokines TNF-α, IL-1β, IL-6, and IFN-y have been shown to dysregulate the KYN pathway, while CRP is a ubiquitous measure of inflammation.
Change in Plasma Kynurenines | 8 weeks
  Blood samples (10 ml) will be collected by a certified phlebotomist at baseline and 8-weeks (post intervention) for the quantification of plasma kynurenines (ng/ml). Plasma concentrations of the kynurenines tryptophan (TRP), kynurenine (KYN), kynurenic acid (KYNA), and quinolinic acid (QUIN) will be quantified in triplicate via enzyme-linked immunosorbent assay (ImmuSmol, Pessac, France).

CONTACTS AND LOCATIONS:
Overall Officials: David J Allison, PhD., Principal Investigator — Lawson Research Institute
Locations (1):
- Parkwood Institute, St Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No